CLINICAL TRIAL: NCT00506909
Title: Double-Blind, Randomized, Placebo-Controlled, Cross-Over Study of Intranasal Oxytocin Augmentation of Antipsychotic Medication in Schizophrenia Patients
Brief Title: Oxytocin Add on Study for Stable Schizophrenic Patients
Acronym: Oxytocin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Break in funding
Sponsor: David Feifel (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor-Investigator, David Feifel, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Oxytocin Schizophrenia
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia
Keywords: oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1: 20 IU BID for the first week, 40IU BID for the following two weeks, 1 week washout, 3 week placebo trial.
  Interventions: Drug: Oxytocin; Drug: Placebo
- Group 2 (Experimental): Group 2: 3 week placebo trial, 1 week washout, 20 IU BID for the first week, 40IU BID for the following two weeks.
  Interventions: Drug: Oxytocin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 20 IU BID or 40 IU BID
Drug: Placebo — 20 IU BID or 40 IU BID

SUMMARY:
The objective of the study is to compare the efficacy of intranasal oxytocin versus intranasal placebo to improve symptoms in schizophrenia patients who have residual symptoms despite being on adequate treatment with antipsychotic medication.

DETAILED DESCRIPTION:
Schizophrenia patients treated with even the best currently available antipsychotic drugs continue to experience significant symptoms. There is a strong need for better treatments including treatments that can safely be given as adjunct to current antipsychotics in order to improve overall efficacy of treatment.

Oxytocin is a neurohypophyseal peptide best known for its role as a neurohormone involved in parturition and lactation. In addition to these well established peripheral effects, there is a compelling body of converging evidence indicating that oxytocin plays a critical role in the regulation of a number of diverse centrally-mediated behavioral and cognitive processes that are highly relevant to Schizophrenia, including social attachment and memory , (see Argiolas and Gessa 1990; McCarthy and Aaltemus 1997).Furthermore, several lines of research suggest that oxytocin receptors may be an important target for development of novel treatments for schizophrenia. Oxytocin and its receptors exist in several areas of the brain which have been heavily implicated in the pathophysiology of schizophrenia, such as the nucleus accumbens and the hippocampus, (Van Leeuwan et al 1985). Oxytocin administered peripherally inhibits dopamine transmission in the mesolimbic pathway (Sarnyai 1992) et al, 1990). Antipsychotics have been found to elevate the secretion of oxytocin in rats (Uvnas-Moberg et al 1992a) suggesting that endogenous oxytocin may play a role in the therapeutic effects of antipsychotic drugs.

Each subject will be enrolled for 6 week treatment period after a screening phase Study procedure involves weekly clinic visits as an outpatient. Forty patients will be randomly assigned to either 40 IU oxytocin twice daily or vehicle placebo. After 3 weeks, treatments will be crossed over such that subjects that received oxytocin will receive placebo and vice versa. The study ratio is 1:1. Dose of oxytocin is based upon previous studies in humans showing improvement in schizophrenia related changes in behavior and brain function (Kosfeld et al, 2005; Kirsch 2005; Heinrich M 2003).

The total study duration for each individual subject will be approximately 7 weeks, which includes up to 7-day screening period, a baseline (randomization) visit, three week treatment period, 1 week washout, baseline, and three weeks cross over treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women, 18 years of age or older.
2. Meet DSM-IV criteria for Schizophrenia.
3. Women of childbearing potential must test negative for pregnancy at the time of enrollment based on urine pregnancy test and agree to use a reliable method of birth control during the study.
4. Must be on a therapeutic dose of an atypical antipsychotic medication (examples but not limited to Clozapine Olanzapine, Risperidone, Ziprasidone, Aripiprazole, Seroquel) with no major dose changes for at least 4 weeks.
5. A minimum PANSS total score of 55 at screening and baseline and a score of at least 4 (moderate) on the subscale of the PANSS (suspiciousness/persecution) at screening.
6. Have a Clinical Global Impressions-Severity (CGI-S) scale score of at least 4 (moderately ill) at baseline.
7. Must be able to communicate effectively with the investigator and study coordinator and have the ability to provide informed consent.
8. Must be able to use nasal spray.
9. Must demonstrate an acceptable degree of compliance with medication and procedures in the opinion of the investigator.

Exclusion Criteria:

Subjects will be excluded from the study of they meet any of the following criteria:

1. Are pregnant or are breastfeeding (negative pregnancy test at screening).
2. A urine drug screen performed at screening must not show evidence of recent use of drugs of abuse.
3. Any active medical condition that in the opinion of the investigator will interfere with the objectives of the study.
4. Are unsuitable in any way to participate in this study, in the opinion of the investigator.
5. Another current DSM-IV diagnosis other than Schizophrenia.

Permitted:

Subjects on one SSRI, and/or sleep medication (diphenhydramine, zolpidem, zaleplon, or diazepam), at a reasonable dose, as judged by the investigator, is permitted in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Feifel, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Feifel D, Macdonald K, Cobb P, Minassian A. Adjunctive intranasal oxytocin improves verbal memory in people with schizophrenia. Schizophr Res. 2012 Aug;139(1-3):207-10. doi: 10.1016/j.schres.2012.05.018. Epub 2012 Jun 8. PMID 22682705
- [Derived] Feifel D, Macdonald K, Nguyen A, Cobb P, Warlan H, Galangue B, Minassian A, Becker O, Cooper J, Perry W, Lefebvre M, Gonzales J, Hadley A. Adjunctive intranasal oxytocin reduces symptoms in schizophrenia patients. Biol Psychiatry. 2010 Oct 1;68(7):678-80. doi: 10.1016/j.biopsych.2010.04.039. Epub 2010 Jul 7. PMID 20615494

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Period: Overall Study
Arm/Group | All Participants
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Total Score in the Positive and Negative Syndrome Scale (PANSS)
Time Frame: performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: Clinical Global Impression-Severity of Illness
Time Frame: performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Calgary Depression Scale for Schizophrenia
Time Frame: performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Clinical Global Impression-Global Improvement
Time Frame: Performed at Visits 2-8 (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: Global Assessment of Functioning
Time Frame: performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Hamilton Anxiety Scale
Time Frame: performed at each visit (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Peabody Picture Vocabulary Test
Time Frame: Visit 1 only
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Letter Number Sequencing Memory Test
Time Frame: Visits 1, 4, and 8 (every 4 weeks)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Reading Trust in the Eyes Test (RTET)
Time Frame: Visits 1, 4, 5 and 8 (every 4 weeks)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: California Verbal Learning Test-Second Edition
Time Frame: Visits 1, 4, and 8 (every 4 weeks)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Profile of Mood States
Time Frame: Visits 1 and 5 (first visit and 5 weeks later)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Paranoid Thought Scale
Time Frame: Visits 1-8 (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Arizona Sexual Experience Scale (ASEX)
Time Frame: Visits 1-8 (weekly)
Population: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Groups:
- All Participants: The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The PI has left the institution and this study was terminated due to loss of funding. The data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes